CLINICAL TRIAL: NCT02548351
Title: A Phase 3, Double-Blind, Randomized, Long-Term, Placebo-Controlled, Multicenter Study Evaluating the Safety and Efficacy of Obeticholic Acid in Subjects With Nonalcoholic Steatohepatitis
Brief Title: Randomized Global Phase 3 Study to Evaluate the Impact on NASH With Fibrosis of Obeticholic Acid Treatment
Acronym: REGENERATE
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The FDA issued a CRL in response to Intercept's NDA for OCA for the treatment of NASH. Sponsor decided to terminate 747-303 before the planned completion date.
Sponsor: Intercept Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 747-303
Record Dates: First submitted 2015-09-01; First posted 2015-09-14 (Estimated); Results first posted 2024-09-05 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-09

CONDITIONS: Non Alcoholic Steatohepatitis (NASH)
Keywords: Non Alcoholic Steatohepatitis, fatty liver disease, NASH
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease | interventions — obeticholic acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 10 mg Obeticholic Acid (Experimental): 10 mg Obeticholic Acid daily for the remainder of the study
  Interventions: Drug: Obeticholic Acid
- 25 mg Obeticholic Acid (Experimental): 25 mg Obeticholic Acid daily for the remainder of the study
  Interventions: Drug: Obeticholic Acid
- Placebo (Placebo Comparator): One tablet daily for the remainder of the study
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Obeticholic Acid
  Arms: 10 mg Obeticholic Acid; 25 mg Obeticholic Acid
Drug: Placebo
  Arms: Placebo

SUMMARY:
The primary objectives of this study are to evaluate the effect of Obeticholic Acid treatment compared to placebo on 1) histological improvement and 2) liver-related clinical outcomes in patients with non-cirrhotic nonalcoholic steatohepatitis (NASH) with liver fibrosis.

ELIGIBILITY:
Inclusion Criteria:

1. Histologic evidence of NASH upon central read of a liver biopsy obtained no more than 6 months before Day 1 defined by presence of all 3 key histological features of NASH according to NASH CRN criteria.
2. Histologic evidence of fibrosis stage 2 or stage 3 as defined by the NASH CRN scoring of fibrosis, or

   Histologic evidence of fibrosis stage 1a or stage 1b if accompanied by ≥1 of the following risk factors:
   * Obesity (BMI ≥30 kg/m2)
   * Type 2 diabetes diagnosed per 2013 American Diabetes Association criteria
   * ALT >1.5× upper limit of normal (ULN).
3. For subjects with a historical biopsy, is either not taking or is on stable doses of TZDs/glitazones or vitamin E for 6 months before Day 1.
4. Stable body weight.

Exclusion Criteria:

1. Model for End-stage Liver Disease (MELD) score >12
2. ALT ≥10× ULN
3. HbA1c >9.5%
4. Total bilirubin >1.5 mg/dL
5. Evidence of other known forms of known chronic liver disease such as alcoholic liver disease, hepatitis B, hepatitis C, PBC, PSC, autoimmune hepatitis, Wilson disease, iron overload, alpha-1-antitrypsin deficiency, drug-induced liver injury, known or suspected hepatocellular carcinoma (HCC)
6. History of liver transplant, or current placement on a liver transplant list
7. Current or history of significant alcohol consumption
8. Prior or planned ileal resection, or prior or planned bariatric surgery
9. Histological presence of cirrhosis
10. History of biliary diversion
11. Known positivity for human immunodeficiency virus infection.
12. Acute cholecystitis or acute biliary obstruction.
13. BMI >45 kg/m2

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2477 (Actual)
Dates: Start 2015-09-22 (Actual); Primary Completion 2023-09-15 (Actual); Study Completion 2023-09-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sangeeta Sawhney, MD, Study Director — Intercept Pharmaceuticals
Locations (346):
- United States (175):
  - The University of Alabama at Birmingham, Birmingham, Alabama
  - Digestive Health Specialists of the Southeast, Dothan, Alabama
  - Institute for Liver Health DBA Arizona Liver Health, Chandler, Arizona
  - Arizona Liver Health - Glendale, Glendale, Arizona
  - St. Joseph's Hospital and Medical Center, Phoenix, Arizona
  - Mayo Clinic Arizona, Phoenix, Arizona
  - Arizona Liver Clinic - Tucson, Tucson, Arizona
  - Liver Wellness Center, Little Rock, Arkansas
  - Arkansas Gastroenterology, North Little Rock, Arkansas
  - GW Research Inc., Chula Vista, California
  - Precision Research Institute, Chula Vista, California
  - Southern California Research Center, Coronado, California
  - Citrus Valley Gastroenterology, Covina, California
  - TriWest Research Associates, LLC, El Cajon, California
  - UCSF Fresno, Clinical Research Center, Fresno, California
  - Fresno Clinical Research Center, Fresno, California
  - Scripps Clinic, La Jolla, California
  - University of California, San Diego, La Jolla, California
  - Keck Medical Center of USC, Los Angeles, California
  - Cedars-Sinai Medical Center, Los Angeles, California
  - National Research Institute, Wilshire, Los Angeles, California
  - Gastrointestinal Biosciences, Los Angeles, California
  - Veteran Affairs Great Los Angeles Healthcare System, Los Angeles, California
  - Stanford University, Palo Alto, California
  - Inland Empire Liver Foundation, Rialto, California
  - University of California Davis Medical Center, Sacramento, California
  - eStudy Site, San Diego, California
  - Medical Associates Research Group, San Diego, California
  - Kaiser Permanente, San Diego, California
  - California Pacific Medical Center (CPMC), San Francisco, California
  - UCSF/ San Francisco General Hospital, San Francisco, California
  - Quest Clinical Research, San Francisco, California
  - University of California, San Francisco, San Francisco, California
  - Silicon Valley Research Institute, San Jose, California
  - University of Colorado Denver and Hospital, Aurora, Colorado
  - South Denver Gastroenterology, PC, Englewood, Colorado
  - Western States Clinical Research, Inc., Wheat Ridge, Colorado
  - Yale University School of Medicine, New Haven, Connecticut
  - Integrity Clinical Research, LLC, Doral, Florida
  - UF Hepatology Research at CTRB, Gainesville, Florida
  - Nature Coast Clinical Research, Inverness, Florida
  - UF Health Jacksonville-Gastroenterology Emerson, Jacksonville, Florida
  - Mayo Clinic, Jacksonville, Florida
  - Florida Digestive Health Specialist Research Institute, Lakewood Rch, Florida
  - Sunrise Medical Research, Inc., Lauderdale Lakes, Florida
  - Meridien Research, Maitland, Florida
  - Bruce W. Carter Miami VA Medical Center, Miami, Florida
  - Schiff Center for Liver Diseases, Miami, Florida
  - ProLive Medical Research, Miami, Florida
  - Janus Clinical Research, Inc., Miami, Florida
  - Sensible Healthcare, LLC, Ocoee, Florida
  - Florida Hospital Transplant Institute, Orlando, Florida
  - South Florida Center of Gastroenterology, P.A., Wellington, Florida
  - Florida Medical Clinic, P.A., Zephyrhills, Florida
  - Summit Clinical Research, LLC, Athens, Georgia
  - Digestive Healthcare of Georgia, Atlanta, Georgia
  - Piedmont Atlanta Hospital, Atlanta, Georgia
  - The Emory Clinic (TEC), Atlanta, Georgia
  - Gastrointestinal Specialists of Georgia, Marietta, Georgia
  - The Queen's Medical Center - Liver Center, Honolulu, Hawaii
  - Grand Teton Research Group, Idaho Falls, Idaho
  - Northwestern University, Feinberg School of Medicine, Chicago, Illinois
  - The University of Chicago Medical Center, Chicago, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Indiana University Health University Hospital, Indianapolis, Indiana
  - Indianapolis Gastroenterology & Hepatology, Indianapolis, Indiana
  - The University of Kansas Medical Center, Kansas City, Kansas
  - The Medical Center of Bowling Green, Bowling Green, Kentucky
  - University of Kentucky Chandler Medical Center, Lexington, Kentucky
  - University of Louisville Medical, Clinical Trials Unit, Louisville, Kentucky
  - Tulane Medical Center, New Orleans, Louisiana
  - Ochsner Clinic Foundation, New Orleans, Louisiana
  - Louisiana Research Center, LLC, Shreveport, Louisiana
  - Investigative Clinical Research, Annapolis, Maryland
  - Mercy Medical Center, Baltimore, Maryland
  - Johns Hopkins Hospital, Baltimore, Maryland
  - Walter Reed National Military Medical Center, Bethesda, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Boston Medical Center, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Lahey Hospital & Medical Center, Burlington, Massachusetts
  - University of Massachusetts Medical School, Worcester, Massachusetts
  - Henry Ford Health System, Detroit, Michigan
  - Gastroenterology Associates of Western Michigan, d.b.a West Michigan Clinical Research, Wyoming, Michigan
  - Huron Gastroenterology Associates/Center for Digestive Care, Ypsilanti, Michigan
  - Minnesota Gastroenterology, Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - Southern Therapy and Advanced Research, LLC, Jackson, Mississippi
  - Kansas City VA Medical Center, Kansas City, Missouri
  - Kansas City Research Institute, Kansas City, Missouri
  - Saint Louis University Gastroenterology & Hepatology, St Louis, Missouri
  - Washington University School of Medicine - Gastroenterology, St Louis, Missouri
  - CHI Health Alegent Creighton Clinic Gastroenterology, Omaha, Nebraska
  - AGA Clinical Research Associates, LLC, Egg Harbor, New Jersey
  - Amici Clinical Research, Martinsville, New Jersey
  - Amici GI - LLC, Martinsville, New Jersey
  - Rutgers University New Jersey Medical School, Newark, New Jersey
  - Saint Joseph's Regional Medical Center, Paterson, New Jersey
  - AccumetRx Clinical research / UGNM, Albuquerque, New Mexico
  - University at Buffalo, Clinical and Translational Research Center, Buffalo, New York
  - Mount Sinai Beth Israel, New York, New York
  - Concorde Medical Group PLLC, New York, New York
  - New York University (NYU) Langone Medical Center, New York, New York
  - Weill Cornell Medical College, New York, New York
  - Icahn School of Medicine at Mt. Sinai, New York, New York
  - Columbia University Medical Center, New York, New York
  - University of Rochester Medical Center, Rochester, New York
  - Montefiore Medical Center, The Bronx, New York
  - Asheville Gastroenterology Associates, PA, Asheville, North Carolina
  - University of North Carolina at Chapel Hill, School of Medicine, Chapel Hill, North Carolina
  - Center for Liver Disease, Charlotte, North Carolina
  - Charlotte Gastroenterology & Hepatology, Charlotte, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Cumberland Research Associates, LLC, Fayetteville, North Carolina
  - Carolinas Center for Liver Disease/Carolinas HeatlhCare System, Huntersville, North Carolina
  - Digestive Health Specialists, PA, Winston-Salem, North Carolina
  - Consultants for Clinical Research, Cincinnati, Ohio
  - University of Cincinnati, Cincinnati, Ohio
  - University Hospitals Case Medical Center, Cleveland, Ohio
  - MetroHealth Medical Center, Cleveland, Ohio
  - The Ohio State University Wexner Medical Center, Columbus, Ohio
  - INTEGRIS Baptist Medical Center, Oklahoma City, Oklahoma
  - Doylestown Health Gastroenterology, Doylestown, Pennsylvania
  - Hillmont GI, pc, Flourtown, Pennsylvania
  - The Pennsylvania State University and The Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Hillmont G.I. - Lansdale Office, Lansdale, Pennsylvania
  - Drexel University, Philadelphia, Pennsylvania
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - Einstein Healthcare Network, Philadelphia, Pennsylvania
  - UPMC, Pittsburgh, Pennsylvania
  - University Gastroenterology, Providence, Rhode Island
  - Prisma Health- Upstate Gastroenterology and Liver Center, Greenville, South Carolina
  - Rapid City Medical Center, Rapid City, South Dakota
  - WR-Clinsearch, LLC, Chattanooga, Tennessee
  - Gastro One, Germantown, Tennessee
  - Associates in Gastroenterology, PLC, Hermitage, Tennessee
  - Clinical Research Solutions, Jackson, Tennessee
  - East Tennesse Research Institute, Johnson City, Tennessee
  - Methodist Healthcare, University Hospital, Memphis, Tennessee
  - Nashville Gastrointestinal Specialists, Nashville, Tennessee
  - Quality Medical Research, PLLC, Nashville, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Texas Clinical Research Institute, Arlington, Texas
  - The Liver Institute at Methodist Dallas Medical Center, Dallas, Texas
  - Liver Center of Texas, Dallas, Texas
  - Texas Digestive Disease Consultants, Dallas, Texas
  - UT Southwestern Medical Center, Dallas, Texas
  - MedResearch, Inc., El Paso, Texas
  - Brooke Army Medical Center, Fort Sam Houston, Texas
  - Baylor Scott & White All Saints Medical Center, Fort Worth, Texas
  - Texas Digestive Disease Consultants, Fort Worth, Texas
  - Baylor College of Medicine Ben Taub General Hospital, Houston, Texas
  - Baylor College of Medicine, Houston, Texas
  - Houston Methodist Hospital, Houston, Texas
  - Liver Associates of Texas, P.A., Houston, Texas
  - The University of Texas Health Science Center at Houston-Medical School IM-Division of Gastroenterology, Hepatology & Nutrition, Houston, Texas
  - Centex Studies, Inc., Houston, Texas
  - Centex Studies, Inc., McAllen, Texas
  - American Research Corporation at the Texas Liver Institute, San Antonio, Texas
  - Gastroenterology Consultants of San Antonio, San Antonio, Texas
  - Texas Digestive Disease Consultants - San Marcos, San Marcos, Texas
  - University of Utah Hospital, Salt Lake City, Utah
  - The University of Vermont Medical Center - Smith 2, Burlington, Vermont
  - University of Virginia Health System, Charlottesville, Virginia
  - Inova Fairfax Medical Campus, Falls Church, Virginia
  - Digestive and Liver Disease Specialists, Norfolk, Virginia
  - Bon Secours St. Mary's Hospital, Richmond, Virginia
  - McGuire DVAMC GI, Richmond, Virginia
  - Virginia Commonwealth University Clinical Research Services Unit (CRSU), Richmond, Virginia
  - Virginia Mason - Seattle Medical Center, Seattle, Washington
  - Swedish Organ Transplant and Liver Center, Seattle, Washington
  - Liver Institute Northwest, Seattle, Washington
  - University of Washington Medical Center, Seattle, Washington
  - University of Wisconsin Hospital & Clinics, Madison, Wisconsin
- Australia (12):
  - Royal Adelaide Hospital Gastroenterology and Hepatology Dept., Adelaide
  - Flinders Medical Centre, Bedford Park
  - AW Morrow Gastroenterology and Liver Centre Royal Prince Alfred Hospital, Camperdown
  - Monash Health - Monash Medical Centre, Clayton
  - Gallipoli Medical Research Foundation, Greenslopes
  - Austin Hospital, Heidelberg
  - Royal Brisbane and Women's Hospital, Herston
  - Nepean Hospital, Kingswood
  - The Alfred Hospital, Department of Gastroenterology, Melbourne
  - Fiona Stanley Hospital, Murdoch
  - The Royal Melbourne Hospital, Parkville
  - Westmead Hospital, Westmead
- Austria (5):
  - Universitätsklinik für Innere Medizin I Innsbruck, Innsbruck
  - Klinikum Klagenfurt am Wörthersee, Klagenfurt
  - Ordensklinikum Linz GmbH, Linz
  - Uniklinikum Salzburg, Salzburg
  - Medizinische Universität Wien, Vienna
- Belgium (8):
  - UZ Antwerpen, Edegem, Antwerpen
  - ULB Hȏpital Erasme - Gastroenterology, Brussels, Brabant
  - UZ Leuven Campus Gathuisberg Hepatology Department, Leuven, Vlaams-Brabant
  - AZ Sint-Jan Brugge Oostende, Bruges
  - UCL Saint-Luc - Hepatology Department, Brussels
  - Ziekenhuis Oost-Limburg (ZOL), Genk
  - UZ Gent Gastroenterology Department, Ghent
  - AZ Nikolaas, Sint-Niklaas
- Canada (13):
  - London Health Sciences Centre University Hospital, London, Ontario
  - University of Calgary Liver Unit, Calgary
  - GI Research, Edmonton
  - University of Alberta, Edmonton
  - Centre de Recherche du Centre Hospitalier de l'Universite de Montreal, Montreal
  - The Research Institute of the McGill University Health Centre, Montreal
  - Toronto Center for Liver Disease, Toronto
  - Toronto Liver Centre, Toronto
  - LAIR Centre, Vancouver
  - Gordon and Leslie Diamond Health Care Centre, Vancouver
  - GIRI - GI Research Institute, Vancouver
  - PerCuro Clinical Research Ltd., Victoria
  - John Buhler Research Centre, Winnipeg
- Denmark (4):
  - Aalborg University Hospital, Aalborg
  - Aarhus University Hospital Medicinsk Hepatogastroenterologisk Afdeling, Aarhus
  - Copenhagen University Hospital Hvidovre, Hvidovre
  - Odense University Hospital, Odense
- Finland (2):
  - Helsinki University Hospital, Helsinki
  - Turku University Hospital, Turku
- France (19):
  - CHU Amiens Picardie, Amiens
  - CHU Angers-Service d'Hepato-Gastroenterologie, Angers
  - Centre hospitalier Pierre Oudot, Bourgoin
  - CHU Beaujon-Service d'Hépatologie, Clichy
  - Hôpital Henri Mondor - Service d'hépatologie, Créteil
  - CHU Grenoble, Grenoble
  - CHRU Hôpital Claude Huriez, Lille
  - Hôpital de la Croix Rousse, Lyon
  - Hôpital Saint Joseph, Marseille
  - Hôpital de l'Archet II-CHU Nice, Nice
  - Service d'Hepato-Gastroenterologie CHR Orleans - La Source, Orléans
  - Hospital Saint Antoine Department of Hepatology, Paris
  - Hôpital de la Pitié Salpétrère, Paris
  - Hôpital Cochin, Paris
  - Hopital Haut-Lévêque-Hépatogastroentérologie-Bât USN, Pessac
  - CHU de Rouen, Rouen
  - CHU Toulouse - Hopital de Purpan, Toulouse
  - CHU de Nancy - Hôpital de Brabois adultes, Vandœuvre-lès-Nancy
  - Hopital Paul Brousse, Villejuif
- Germany (17):
  - Universitätsklinikum Heidelberg Medizinischen Klinik IV Gastroenterologie und Hepatologie, Heidelberg, Baden-Wurttemberg
  - Friedrich-Alexander-Universität Erlangen Medizinische Klinik 1, Erlangen, Bavaria
  - Universitätsmedizin Mainz, I. Med. Klinik und Poliklinik, Mainz, Rhineland-Palatinate
  - Universitätsklinikum Leipzig Klinik für Gastroenterologie und Rheumatologie-Sektion Hepatologie, Leipzig, Saxony
  - Universitatsklinikum Aachen, RWTH Aachen, Medizinische Klinik III, Aachen
  - Charite Universitätsmedizin Campus Virchow, Berlin
  - St. Josef-Hospital, Ruhr University Bochum, Bochum
  - University Hosptial Cologne Clinics for Gastroenterology and Hepatology, Cologne
  - University Hospital Essen, Essen
  - Katholische Kliniken Ruhrhalbinsel GmbH, Essen
  - Universitätsklinikum Hamburg- Eppendorf, Hamburg
  - Medizinische Hochschule Hannover, Hanover
  - Gastroenterologische Gemeinschaftspraxis, Herne
  - Hepato-Gastroenterology Center Kiel, Kiel
  - EUGASTRO GmbH, Leipzig
  - Krankenhaus Barmherzige Bruder Innere Medizin I - Gastroenterologie, Munich
  - Universitätsklinikum Würzburg, Würzburg
- Hungary (3):
  - Egyesitett Szent Istvan és Szent Laszlo, Budapest
  - Pecsi Tudomanyegyetem Klinikai Kozpont, I. sz, Budapest
  - Kenezy Gyula Korhaz es Rendelointezet, Debrecen
- Israel (10):
  - Soroka Medical Center Division of Internal Medicine, Beersheba
  - Rambam Medical Center Center for Liver diseases, Haifa
  - Carmel Medical Center, Haifa
  - Shaarei Zedek Medical Center, Jerusalem
  - Hadassah Ein Kerem MC, Jerusalem
  - West Galilee Hospital, Nahariya
  - Holy Family Medical Center, Nazareth
  - Rabin Medical Center, Liver Institute, Petah Tikva
  - Sheba Medical Center, Ramat Gan
  - Sourasky Tel-Aviv Medical Center, Tel Aviv
- Italy (12):
  - Universita di Bologna - DIMEC, Bologna
  - University di Bologna - Dipartimento di Scienze Mediche e Chirurgiche - DIMEC, Bologna
  - Ospedale san Giuseppe - Multimedica, Milan
  - Fondazione IRCCS Ca Granda Ospedale, Milan
  - Azienda Socio-Sanitaria Territoriale (ASST) Santi Paolo e Carlo, Milan
  - Fondazione IRCCS Ca Grande Ospedale, Milan
  - AOU di Modena Ospedale Civile, Modena
  - Azienda Ospedaliera Universitaria Policlinico, Napoli
  - Policlinico Paolo Giaccone di Palermo, Palermo
  - Policlinico University Campus Biomedico, Rome
  - Istituto Clinico Humanitas, Rozzano
  - A.O.U. Città della Salute e della Scienza di Torino, Torino
- New Zealand (2):
  - NZ Liver Transplant Unit, Grafton, Auckland
  - Middlemore Hospital, Auckland
- Poland (5):
  - Centrum Badan Klinicznych PI-House Sp. z o.o., Gdansk
  - Uniwersyteckie Centrum Kliniczne im. Prof K. Gibinskiego Slaskiego Uniwersytetu Medycznego w Katowicach, Katowice
  - Wojewodzki Specjalistyczny Szpital im. Dr WI. Bieganskiego, Lodz
  - Samodzielny Publiczny Szpital Kliniczny Nr 1, Lublin
  - Centrum Badan Klinicznych Piotr Napora, Wroclaw
- Portugal (5):
  - Centro Hospitalar do Baixo Vouga, E.P.E., Aveiro
  - Ulsba, Epe, Beja
  - Hospital da Senhora da Oliveira - Guimarães, Guimarães
  - Centro Hospitalar Lisboa Ocidental, Lisbon
  - Centro Hospitalar de Lisboa Norte, EPE - Hosp. de Santa Maria, Lisbon
- Puerto Rico (3):
  - Klinical Investigations Group, LLC, San Juan
  - Ave Ponce De Leon #715, San Juan
  - Fundacion de Investigacion, San Juan
- Serbia (3):
  - University Medical Centar Zvezdara, Belgrade
  - Clinical Hospital Center Bezanijska Kosa, Belgrade
  - Clinical Center Nis, Niš
- Spain (19):
  - Hospital Universitari Son Espases, Palma de Mallorca, Balearic Islands
  - Hospital Universitario Puerta de Hierro Majadahonda, Majadahonda, Madrid
  - Hospital Universitario Fundación Alcorcon, Alcorcón
  - Hospital General y Universitario de Alicante, Alicante
  - Hospital del Mar Gastroenterology Department, Barcelona
  - Hospital Universitario Vall d'Hebron, Barcelona
  - Hospital Clinic(o) de Barcelona, Barcelona
  - Hospital Universitario Donostia, Donostia / San Sebastian
  - Complejo Asistencial Universitario de Leon, León
  - Hospital Universitario Ramón y Cajal, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital (Universitario) Virgen de la Victoria, Málaga
  - Hospital (Universitario) Marqués de Valdecilla, Santander
  - Hospital Clinico Universitario de Santiago, Santiago de Compostela
  - Hospital Universitario Virgen del Rocio, Seville
  - Hospital Clinico Universitario de Valencia, Valencia
  - Consorcio Hospital General Universitario, Valencia
  - Hospital Universitario La Fe., Valencia
  - Hospital Universitario Miguel Servet, Zaragoza
- Sweden (3):
  - Sahlgrenska University Hospital, Gothenburg
  - Universitetsjukhuset Linkoping, Linköping
  - Karolinska University Hospital, Stockholm
- Switzerland (4):
  - UVCM Hepatologie, Bern
  - Epatocentro Ticino, Lugano
  - Hospital of St. Gallen, Sankt Gallen
  - University Clinic of Gastroenterology & Hepatology, Zurich
- United Kingdom (22):
  - Royal Cornwall Hospital, Truro, Cornwall
  - Royal Bournemouth Hospital, Bournemouth, Dorset
  - Queen Alexandra Hospital, Portsmouth, Hampshire
  - Norfolk and Norwich University Hospitals, Norwich, Norfolk
  - John Radcliffe Hospital, Headington, Oxford
  - Royal Surrey NHS Foundation Trust, Guildford, Surrey
  - Institute of Biomedical Research, Birmingham
  - Bradford Royal Infirmary, Bradford
  - University Hospital Bristol NHS Foundation Trust, Bristol
  - Cambridge University Hospital, Cambridge
  - University Hospitals Coventry & Warwickshire, Coventry
  - Glasgow Royal Infirmary, NHS Greater, Glasgow
  - Gastroenterology Department Hull Royal Infirmary, Hull
  - University Hospital Aintree, Liverpool
  - Royal London Hospital, London
  - Institute for Liver and Digestive Health, London
  - Guy's and St. Thomas NHS Foundation Trust, London
  - St. Mary's Hospital, London
  - Central Manchester University Hospital NHS Foundation Trust Manchester Royal Infirmary, Manchester
  - The Newcastle Upon Tyne Hospitals NHS Foundation Trust, Newcastle upon Tyne
  - Nottingham Digestive Diseases and Biomedical Research Unit, Nottingham
  - Derriford Hospital, Plymouth

REFERENCES:
- [Derived] Sanyal AJ, Loomba R, Anstee QM, Ratziu V, Kowdley KV, Rinella ME, Harrison SA, Resnick MB, Capozza T, Sawhney S, Shelat N, Younossi ZM. Utility of pathologist panels for achieving consensus in NASH histologic scoring in clinical trials: Data from a phase 3 study. Hepatol Commun. 2023 Dec 22;8(1):e0325. doi: 10.1097/HC9.0000000000000325. eCollection 2024 Jan 1. PMID 38126958
- [Derived] Rinella ME, Dufour JF, Anstee QM, Goodman Z, Younossi Z, Harrison SA, Loomba R, Sanyal AJ, Bonacci M, Trylesinski A, Natha M, Shringarpure R, Granston T, Venugopal A, Ratziu V. Non-invasive evaluation of response to obeticholic acid in patients with NASH: Results from the REGENERATE study. J Hepatol. 2022 Mar;76(3):536-548. doi: 10.1016/j.jhep.2021.10.029. Epub 2021 Nov 15. PMID 34793868
- [Derived] Younossi ZM, Stepanova M, Nader F, Loomba R, Anstee QM, Ratziu V, Harrison S, Sanyal AJ, Schattenberg JM, Barritt AS, Noureddin M, Bonacci M, Cawkwell G, Wong B, Rinella M; RandomizEd Global Phase 3 Study to Evaluate the Impact on NASH with FibRosis of Obeticholic Acid TreatmEnt (REGENERATE) Study Investigators. Obeticholic Acid Impact on Quality of Life in Patients With Nonalcoholic Steatohepatitis: REGENERATE 18-Month Interim Analysis. Clin Gastroenterol Hepatol. 2022 Sep;20(9):2050-2058.e12. doi: 10.1016/j.cgh.2021.07.020. Epub 2021 Jul 15. PMID 34274514
- [Derived] Younossi ZM, Ratziu V, Loomba R, Rinella M, Anstee QM, Goodman Z, Bedossa P, Geier A, Beckebaum S, Newsome PN, Sheridan D, Sheikh MY, Trotter J, Knapple W, Lawitz E, Abdelmalek MF, Kowdley KV, Montano-Loza AJ, Boursier J, Mathurin P, Bugianesi E, Mazzella G, Olveira A, Cortez-Pinto H, Graupera I, Orr D, Gluud LL, Dufour JF, Shapiro D, Campagna J, Zaru L, MacConell L, Shringarpure R, Harrison S, Sanyal AJ; REGENERATE Study Investigators. Obeticholic acid for the treatment of non-alcoholic steatohepatitis: interim analysis from a multicentre, randomised, placebo-controlled phase 3 trial. Lancet. 2019 Dec 14;394(10215):2184-2196. doi: 10.1016/S0140-6736(19)33041-7. Epub 2019 Dec 5. PMID 31813633
- [Derived] Ratziu V, Sanyal AJ, Loomba R, Rinella M, Harrison S, Anstee QM, Goodman Z, Bedossa P, MacConell L, Shringarpure R, Shah A, Younossi Z. REGENERATE: Design of a pivotal, randomised, phase 3 study evaluating the safety and efficacy of obeticholic acid in patients with fibrosis due to nonalcoholic steatohepatitis. Contemp Clin Trials. 2019 Sep;84:105803. doi: 10.1016/j.cct.2019.06.017. Epub 2019 Jun 29. PMID 31260793

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a phase 3, double-blind, randomized, long-term, placebo-controlled, multicenter study evaluating the safety and efficacy of Obeticholic Acid (OCA) in Participants with Nonalcoholic Steatohepatitis (NASH).
Pre-assignment Details: The study was conducted at approximately 350 investigational sites globally.
Groups:
- OCA 10 Milligrams (mg): Participants were randomized to receive OCA 10 mg once daily orally with water.
- OCA 25 mg: Participants were randomized to receive OCA 25 mg once daily orally with water.
- Placebo: Participants were randomized to receive matching placebo once daily orally with water.
Period: Overall Study
Arm/Group | OCA 10 Milligrams (mg) | OCA 25 mg | Placebo
Started | 825 | 827 | 825
Completed | 0 | 0 | 0
Not Completed | 825 | 827 | 825
Not completed — Withdrawal by Subject | 149 | 154 | 152
Not completed — Death | 11 | 15 | 12
Not completed — Adverse Event | 22 | 56 | 36
Not completed — Study Terminated by Sponsor | 549 | 509 | 528
Not completed — Site Closure | 14 | 5 | 7
Not completed — Non-compliance with Study Drug | 4 | 2 | 0
Not completed — Protocol Violation | 2 | 1 | 2
Not completed — Physician Decision | 11 | 18 | 11
Not completed — Lost to Follow-up | 43 | 50 | 57
Not completed — Other | 19 | 16 | 20
Not completed — Missing | 1 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | OCA 10 Milligrams (mg) | OCA 25 mg | Placebo | Total
Number analyzed (Participants) | 825 | 827 | 825 | 2477
Age, Continuous [Mean (Standard Deviation); unit: Years] | 55.3 (10.76) | 55.3 (11.71) | 54.4 (11.21) | 55.3 (11.24)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 475 | 494 | 478 | 1447
  Male | 350 | 333 | 347 | 1030
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 129 | 149 | 147 | 425
  Not Hispanic or Latino | 620 | 594 | 592 | 1806
  Unknown or Not Reported | 76 | 84 | 86 | 246
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 5 | 8 | 6 | 19
  Asian | 47 | 43 | 29 | 119
  Native Hawaiian or Other Pacific Islander | 4 | 4 | 2 | 10
  Black or African American | 14 | 20 | 12 | 46
  White | 679 | 674 | 685 | 2038
  More than one race | 4 | 3 | 7 | 14
  Unknown or Not Reported | 72 | 75 | 84 | 231

OUTCOME MEASURES:

1. Primary Outcome: Time to the First Adjudicated Event for Clinical Outcome Composite Endpoint: Percentage of Participants With an Event
Description: All potential liver-related clinical outcomes that occurred after administration of first dose of investigational product were reviewed and adjudicated by blinded, independent Hepatic Outcomes Committee(HOC). Adjudicated results were used to assess effect of OCA, compared to placebo in conjunction with established local standard of care, on clinical outcomes in participants with NASH as measured by time to first occurrence of any of following adjudicated events, derived as a composite event endpoint of death(all-cause), liver transplant, Model of End-stage Liver Disease(MELD)≥15 Score, hospitalization(defined by a stay of 24 hours or greater) for onset of: variceal bleed, hepatic encephalopathy(defined by a West Haven score of ≥2), and spontaneous bacterial peritonitis(confirmed by diagnostic paracentesis), ascites secondary to cirrhosis requiring medical intervention, and histological progression to Cirrhosis. Clinical events distribution was estimated using Kaplan-Meier methodology.
Time Frame: Up to 7 years
Population: Intent-to-Treat (ITT) Population comprised of all randomized participants with fibrosis stage 2 or stage 3 who receive at least 1 dose of investigational product.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | OCA 10 Milligrams (mg) | OCA 25 mg | Placebo
Number analyzed (Participants) | 729 | 730 | 728
Percentage of participants | 15.8 [13.2 to 18.6] | 14.7 [12.2 to 17.4] | 18.8 [16.0 to 21.9]
Statistical Analysis 1: Comparison: OCA 10 Milligrams (mg) vs Placebo; Test type: Other; p = 0.1028, Log Rank; Hazard Ratio (HR) = 0.814, 95% CI 2-sided [0.635 to 1.043]
Statistical Analysis 2: Comparison: OCA 25 mg vs Placebo; Test type: Other; p = 0.0444, Log Rank; Hazard Ratio (HR) = 0.772, 95% CI 2-sided [0.600 to 0.994]

2. Secondary Outcome: Percentage of Responders With Improvement of Fibrosis by at Least One Stage With no Worsening of NASH Using Consensus Read Method of Scheduled Liver Biopsies
Description: Fibrosis stage was evaluated by NASH Clinical Research Network (CRN) Fibrosis Staging System as follows: Stage 0: No fibrosis, Stage 1: Perisinusoidal/periportal fibrosis, Stage 1A: Mild, zone 3, perisinusoidal fibrosis, Stage 1B: Moderate, zone 3, perisinusoidal fibrosis, Stage 1C: Portal/periportal fibrosis, Stage 2: Perisinusoidal and portal/periportal fibrosis, Stage 3: Bridging fibrosis and Stage 4: Cirrhosis. No worsening of NASH was defined as no worsening of hepatocellular ballooning, no worsening of lobular inflammation, and no worsening of steatosis. Responders are defined as participants who did not discontinue treatment due to Adverse event (AE) or did not die and had evaluable post-Baseline biopsy assessment. Mantel-Haenszel method is used to construct the confidence intervals.
Time Frame: Up to 7 years
Population: ITT Population.
Measure: Number; unit: Percentage of participants
Arm/Group | OCA 10 Milligrams (mg) | OCA 25 mg | Placebo
Number analyzed (Participants) | 729 | 730 | 728
Percentage of participants | 17.1 | 19.5 | 10.0
Statistical Analysis 1: Comparison: OCA 10 Milligrams (mg) vs Placebo; Test type: Other; p < 0.0001, Cochran-Mantel-Haenszel; Difference in percentages = 7.1, 95% CI 2-sided [3.6 to 10.6]
Statistical Analysis 2: Comparison: OCA 25 mg vs Placebo; Test type: Other; p < 0.0001, Cochran-Mantel-Haenszel; Treatment difference = 9.4, 95% CI 2-sided [5.8 to 13.0]

3. Secondary Outcome: Percentage of Participants Who Showed Improvement in Fibrosis by at Least 1 Stage and/or Resolution of NASH Without Worsening of Either Using Consensus Read Method
Description: Fibrosis stage was evaluated by NASH Clinical Research Network(CRN) Fibrosis Staging System as follows: Stage 0:No fibrosis, Stage 1:Perisinusoidal/periportal fibrosis, Stage 1A:Mild, zone 3, perisinusoidal fibrosis, Stage 1B:Moderate, zone3, perisinusoidal fibrosis, Stage 1C:Portal/periportal fibrosis, Stage 2:Perisinusoidal and portal/periportal fibrosis, Stage 3:Bridging fibrosis and Stage 4:Cirrhosis. Resolution of NASH (Nonalcoholic Steatohepatitis) is defined as absence of fatty liver disease, or presence of simple or isolated steatosis without steatohepatitis, with a NAS(NAFLD Activity Score) of 0 for ballooning and 0 to 1 for inflammation. NAS ranges from 0-12; 0: no features of fatty liver disease and 12: highest degree of fatty liver disease. Higher signify worse symptoms. Responders are who did not discontinue treatment due to Adverse event(AE) or did not die and had evaluable post-Baseline biopsy assessment. Mantel-Haenszel method is used to construct confidence intervals.
Time Frame: Up to 7 years
Population: ITT Population.
Measure: Number; unit: Percentage of participants
Arm/Group | OCA 10 Milligrams (mg) | OCA 25 mg | Placebo
Number analyzed (Participants) | 729 | 730 | 728
Percentage of participants | 18.5 | 20.8 | 11.8
Statistical Analysis 1: Comparison: OCA 10 Milligrams (mg) vs Placebo; Test type: Other; p = 0.0004, Cochran-Mantel-Haenszel; Treatment difference = 6.7, 95% CI 2-sided [3.0 to 10.4]
Statistical Analysis 2: Comparison: OCA 25 mg vs Placebo; Test type: Other; p < 0.0001, Cochran-Mantel-Haenszel; Treatment difference = 9.0, 95% CI 2-sided [5.2 to 12.8]

4. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs)
Description: An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of a study intervention, whether or not considered related to the study intervention. A TEAE was defined as any AE that either newly appeared, increased in frequency, or worsened in severity following treatment up to 30 days from last dose of permanent investigational product discontinuation. Serious AE (SAE) was defined as any AE resulting in death, immediate risk of death, inpatient hospitalization or prolongation of existing hospitalization, persistent or significant disability/incapacity, or a congenital/anomaly/birth defect, or any other medically important event.
Time Frame: Up to 7 years
Population: Safety Population comprised all randomized participants, all fibrosis stages, who receive at least 1 dose of investigational product (OCA or placebo).
Measure: Count of Participants; unit: Participants
Arm/Group | OCA 10 Milligrams (mg) | OCA 25 mg | Placebo
Number analyzed (Participants) | 825 | 827 | 825
Participants
  TEAEs | 798 | 813 | 781
  SAEs | 273 | 276 | 248

ADVERSE EVENTS:
Time Frame: Up to 7 years
Description: Treatment emergent adverse events and serious adverse events were collected in the Safety Population. Safety Population comprises of participants who received at least one dose of study treatment.
Arm/Group | OCA 10 Milligrams (mg) | OCA 25 mg | Placebo
All-Cause Mortality (participants affected / at risk) | 14/825 | 19/827 | 14/825
Serious Adverse Events (participants affected / at risk) | 273/825 | 276/827 | 248/825
Other Adverse Events (participants affected / at risk) | 798/825 | 813/827 | 781/825
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | OCA 10 Milligrams (mg) (N=825) | OCA 25 mg (N=827) | Placebo (N=825)
Anaemia (Blood and lymphatic system disorders) | 4 | 2 | 3
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 0
Pancytopenia (Blood and lymphatic system disorders) | 0 | 0 | 1
Polycythaemia (Blood and lymphatic system disorders) | 1 | 0 | 0
Splenic lesion (Blood and lymphatic system disorders) | 1 | 0 | 0
Acute coronary syndrome (Cardiac disorders) | 1 | 1 | 1
Acute myocardial infarction (Cardiac disorders) | 4 | 7 | 4
Angina pectoris (Cardiac disorders) | 4 | 6 | 2
Angina unstable (Cardiac disorders) | 2 | 2 | 2
Arteriosclerosis coronary artery (Cardiac disorders) | 0 | 0 | 1
Atrial fibrillation (Cardiac disorders) | 8 | 5 | 4
Atrial flutter (Cardiac disorders) | 1 | 1 | 0
Atrioventricular block (Cardiac disorders) | 0 | 0 | 1
Cardiac arrest (Cardiac disorders) | 0 | 1 | 2
Cardiac failure (Cardiac disorders) | 0 | 2 | 1
Cardiac failure congestive (Cardiac disorders) | 1 | 2 | 2
Cardio-respiratory arrest (Cardiac disorders) | 0 | 1 | 0
Cardio-respiratory distress (Cardiac disorders) | 0 | 1 | 0
Congestive cardiomyopathy (Cardiac disorders) | 1 | 0 | 0
Cor pulmonale (Cardiac disorders) | 1 | 0 | 0
Coronary artery disease (Cardiac disorders) | 5 | 4 | 7
Coronary artery occlusion (Cardiac disorders) | 0 | 0 | 1
Coronary artery stenosis (Cardiac disorders) | 2 | 1 | 1
Hypertensive heart disease (Cardiac disorders) | 1 | 0 | 0
Mitral valve incompetence (Cardiac disorders) | 0 | 0 | 1
Myocardial infarction (Cardiac disorders) | 1 | 3 | 0
Myocardial ischaemia (Cardiac disorders) | 4 | 0 | 0
Palpitations (Cardiac disorders) | 0 | 1 | 1
Pericardial effusion (Cardiac disorders) | 1 | 0 | 0
Pericarditis (Cardiac disorders) | 0 | 2 | 1
Pericarditis constrictive (Cardiac disorders) | 0 | 1 | 0
Sinus tachycardia (Cardiac disorders) | 1 | 0 | 0
Supraventricular tachycardia (Cardiac disorders) | 0 | 1 | 0
Tachycardia (Cardiac disorders) | 0 | 0 | 1
Ventricular tachycardia (Cardiac disorders) | 0 | 1 | 0
Arnold-Chiari malformation (Congenital, familial and genetic disorders) | 1 | 0 | 0
Arteriovenous malformation (Congenital, familial and genetic disorders) | 1 | 0 | 0
Congenital cerebrovascular anomaly (Congenital, familial and genetic disorders) | 0 | 0 | 1
Rathke's cleft cyst (Congenital, familial and genetic disorders) | 0 | 0 | 1
Labyrinthine fistula (Ear and labyrinth disorders) | 0 | 0 | 1
Vertigo (Ear and labyrinth disorders) | 1 | 2 | 2
Vertigo positional (Ear and labyrinth disorders) | 1 | 0 | 1
Adrenal haematoma (Endocrine disorders) | 1 | 0 | 0
Goitre (Endocrine disorders) | 1 | 0 | 0
Pituitary-dependent Cushing's syndrome (Endocrine disorders) | 0 | 1 | 0
Thyroid mass (Endocrine disorders) | 0 | 0 | 1
Thyroiditis subacute (Endocrine disorders) | 1 | 0 | 0
Macular fibrosis (Eye disorders) | 0 | 1 | 0
Optic ischaemic neuropathy (Eye disorders) | 0 | 1 | 0
Retinal detachment (Eye disorders) | 0 | 1 | 0
Vision blurred (Eye disorders) | 1 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 1
Abdominal hernia (Gastrointestinal disorders) | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 7 | 4 | 7
Abdominal pain upper (Gastrointestinal disorders) | 2 | 0 | 2
Abdominal wall disorder (Gastrointestinal disorders) | 0 | 0 | 1
Abdominal wall haematoma (Gastrointestinal disorders) | 1 | 0 | 0
Apical granuloma (Gastrointestinal disorders) | 0 | 0 | 1
Appendix disorder (Gastrointestinal disorders) | 1 | 0 | 0
Ascites (Gastrointestinal disorders) | 2 | 2 | 0
Colitis (Gastrointestinal disorders) | 1 | 0 | 1
Colitis ischaemic (Gastrointestinal disorders) | 1 | 1 | 2
Colitis ulcerative (Gastrointestinal disorders) | 0 | 0 | 1
Colonic fistula (Gastrointestinal disorders) | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 3
Diarrhoea (Gastrointestinal disorders) | 0 | 4 | 0
Diverticulum intestinal (Gastrointestinal disorders) | 0 | 0 | 1
Diverticulum intestinal haemorrhagic (Gastrointestinal disorders) | 0 | 0 | 1
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Dyschezia (Gastrointestinal disorders) | 1 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 1 | 1
Enteritis (Gastrointestinal disorders) | 0 | 0 | 1
Enterocolitis (Gastrointestinal disorders) | 0 | 0 | 1
Gastric haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Gastric polyps (Gastrointestinal disorders) | 0 | 0 | 1
Gastric ulcer (Gastrointestinal disorders) | 0 | 1 | 0
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 1 | 2 | 0
Gastritis erosive (Gastrointestinal disorders) | 0 | 1 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 3 | 3 | 2
Haematemesis (Gastrointestinal disorders) | 0 | 1 | 1
Haematochezia (Gastrointestinal disorders) | 0 | 0 | 2
Haemorrhoids (Gastrointestinal disorders) | 0 | 1 | 0
Hiatus hernia (Gastrointestinal disorders) | 0 | 1 | 0
Impaired gastric emptying (Gastrointestinal disorders) | 0 | 3 | 0
Incarcerated umbilical hernia (Gastrointestinal disorders) | 0 | 1 | 0
Inguinal hernia (Gastrointestinal disorders) | 1 | 0 | 0
Intestinal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Intestinal ischaemia (Gastrointestinal disorders) | 1 | 0 | 0
Intestinal obstruction (Gastrointestinal disorders) | 0 | 1 | 2
Intra-abdominal haematoma (Gastrointestinal disorders) | 1 | 0 | 0
Large intestine perforation (Gastrointestinal disorders) | 1 | 0 | 0
Large intestine polyp (Gastrointestinal disorders) | 0 | 0 | 1
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1
Melaena (Gastrointestinal disorders) | 2 | 1 | 0
Nausea (Gastrointestinal disorders) | 2 | 1 | 1
Oesophageal obstruction (Gastrointestinal disorders) | 1 | 0 | 0
Oesophageal varices haemorrhage (Gastrointestinal disorders) | 0 | 2 | 0
Pancreatitis (Gastrointestinal disorders) | 4 | 6 | 1
Pancreatitis acute (Gastrointestinal disorders) | 5 | 1 | 3
Pancreatitis haemorrhagic (Gastrointestinal disorders) | 0 | 0 | 1
Peritoneal haemorrhage (Gastrointestinal disorders) | 1 | 1 | 1
Portal hypertensive gastropathy (Gastrointestinal disorders) | 0 | 1 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 2 | 1 | 1
Retroperitoneal haematoma (Gastrointestinal disorders) | 0 | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 2 | 5 | 5
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 1
Umbilical hernia (Gastrointestinal disorders) | 1 | 1 | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1
Varices oesophageal (Gastrointestinal disorders) | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 2 | 2 | 1
Adverse drug reaction (General disorders) | 0 | 0 | 1
Asthenia (General disorders) | 2 | 2 | 2
Breast complication associated with device (General disorders) | 1 | 0 | 0
Calcinosis (General disorders) | 0 | 1 | 0
Chest discomfort (General disorders) | 0 | 1 | 0
Chest pain (General disorders) | 5 | 8 | 6
Death (General disorders) | 0 | 2 | 0
Device deployment issue (General disorders) | 1 | 0 | 0
Device dislocation (General disorders) | 0 | 1 | 0
Disease progression (General disorders) | 0 | 1 | 0
Dysplasia (General disorders) | 0 | 0 | 1
Impaired healing (General disorders) | 0 | 0 | 1
Mass (General disorders) | 0 | 1 | 0
Non-cardiac chest pain (General disorders) | 3 | 7 | 2
Oedema peripheral (General disorders) | 0 | 1 | 0
Pyrexia (General disorders) | 0 | 3 | 1
Systemic inflammatory response syndrome (General disorders) | 0 | 2 | 0
Vascular stent occlusion (General disorders) | 0 | 1 | 0
Acute hepatic failure (Hepatobiliary disorders) | 0 | 1 | 0
Autoimmune hepatitis (Hepatobiliary disorders) | 0 | 1 | 0
Bile duct obstruction (Hepatobiliary disorders) | 1 | 1 | 0
Bile duct stone (Hepatobiliary disorders) | 3 | 3 | 1
Biliary colic (Hepatobiliary disorders) | 0 | 2 | 1
Biliary tract disorder (Hepatobiliary disorders) | 1 | 0 | 0
Biloma (Hepatobiliary disorders) | 1 | 0 | 0
Cholangitis (Hepatobiliary disorders) | 0 | 2 | 0
Cholangitis acute (Hepatobiliary disorders) | 1 | 0 | 0
Cholecystitis (Hepatobiliary disorders) | 2 | 4 | 4
Cholecystitis acute (Hepatobiliary disorders) | 2 | 9 | 1
Cholecystitis chronic (Hepatobiliary disorders) | 1 | 2 | 0
Cholelithiasis (Hepatobiliary disorders) | 4 | 8 | 4
Cholestasis (Hepatobiliary disorders) | 0 | 1 | 0
Cholestatic liver injury (Hepatobiliary disorders) | 0 | 1 | 0
Chronic hepatic failure (Hepatobiliary disorders) | 0 | 1 | 0
Drug-induced liver injury (Hepatobiliary disorders) | 0 | 3 | 0
Gallbladder perforation (Hepatobiliary disorders) | 0 | 1 | 0
Gallbladder polyp (Hepatobiliary disorders) | 0 | 0 | 1
Hepatic cirrhosis (Hepatobiliary disorders) | 0 | 2 | 1
Hepatic failure (Hepatobiliary disorders) | 1 | 1 | 0
Hepatic haematoma (Hepatobiliary disorders) | 3 | 2 | 2
Hepatic lesion (Hepatobiliary disorders) | 2 | 0 | 0
Hepatitis (Hepatobiliary disorders) | 0 | 1 | 0
Hepatorenal syndrome (Hepatobiliary disorders) | 1 | 1 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 | 2 | 0
Hyperplastic cholecystopathy (Hepatobiliary disorders) | 0 | 1 | 0
Anaphylactic reaction (Immune system disorders) | 0 | 1 | 0
Drug hypersensitivity (Immune system disorders) | 0 | 1 | 1
Hypersensitivity (Immune system disorders) | 0 | 0 | 1
Abscess limb (Infections and infestations) | 1 | 0 | 1
Anal infection (Infections and infestations) | 0 | 1 | 0
Appendicitis (Infections and infestations) | 4 | 4 | 1
Appendicitis perforated (Infections and infestations) | 1 | 0 | 1
Arthritis bacterial (Infections and infestations) | 1 | 0 | 0
Bronchiolitis (Infections and infestations) | 0 | 1 | 0
Bronchitis (Infections and infestations) | 0 | 1 | 1
Cellulitis (Infections and infestations) | 3 | 5 | 6
Cholecystitis infective (Infections and infestations) | 0 | 1 | 0
Chronic sinusitis (Infections and infestations) | 1 | 0 | 0
Clostridium difficile colitis (Infections and infestations) | 0 | 3 | 0
Clostridium difficile infection (Infections and infestations) | 0 | 1 | 0
Coccidioidomycosis (Infections and infestations) | 1 | 0 | 0
Corona virus infection (Infections and infestations) | 6 | 7 | 6
Cystitis (Infections and infestations) | 0 | 3 | 1
Cytomegalovirus mononucleosis (Infections and infestations) | 0 | 1 | 0
Device related infection (Infections and infestations) | 0 | 1 | 0
Diarrhoea infectious (Infections and infestations) | 2 | 1 | 0
Diverticulitis (Infections and infestations) | 3 | 2 | 1
Encephalitis viral (Infections and infestations) | 1 | 0 | 0
Endocarditis bacterial (Infections and infestations) | 1 | 0 | 0
Escherichia sepsis (Infections and infestations) | 1 | 0 | 1
Gangrene (Infections and infestations) | 0 | 0 | 1
Gastroenteritis (Infections and infestations) | 2 | 4 | 2
Gastroenteritis viral (Infections and infestations) | 0 | 1 | 1
Graft infection (Infections and infestations) | 1 | 0 | 0
Groin abscess (Infections and infestations) | 0 | 0 | 1
Helicobacter infection (Infections and infestations) | 0 | 0 | 1
Hepatitis E (Infections and infestations) | 1 | 1 | 0
Histoplasmosis (Infections and infestations) | 1 | 0 | 0
Infection (Infections and infestations) | 1 | 0 | 0
Influenza (Infections and infestations) | 0 | 1 | 0
Joint abscess (Infections and infestations) | 1 | 0 | 0
Kidney infection (Infections and infestations) | 0 | 1 | 1
Liver abscess (Infections and infestations) | 1 | 0 | 0
Localised infection (Infections and infestations) | 0 | 1 | 0
Mastoiditis (Infections and infestations) | 0 | 1 | 1
Medical device site joint infection (Infections and infestations) | 1 | 1 | 0
Osteomyelitis (Infections and infestations) | 1 | 0 | 0
Parotid abscess (Infections and infestations) | 0 | 1 | 0
Pelvic abscess (Infections and infestations) | 0 | 0 | 1
Perirectal abscess (Infections and infestations) | 0 | 1 | 1
Peritonitis (Infections and infestations) | 1 | 1 | 0
Pharyngeal abscess (Infections and infestations) | 1 | 0 | 0
Pneumonia (Infections and infestations) | 5 | 9 | 7
Pneumonia viral (Infections and infestations) | 9 | 10 | 4
Post procedural cellulitis (Infections and infestations) | 0 | 0 | 1
Post procedural infection (Infections and infestations) | 0 | 1 | 0
Post procedural sepsis (Infections and infestations) | 1 | 0 | 0
Postoperative wound infection (Infections and infestations) | 2 | 1 | 0
Pseudomonas infection (Infections and infestations) | 0 | 0 | 1
Pulmonary sepsis (Infections and infestations) | 1 | 0 | 0
Pyelonephritis (Infections and infestations) | 5 | 4 | 3
Rotavirus infection (Infections and infestations) | 0 | 1 | 0
Salmonellosis (Infections and infestations) | 0 | 1 | 0
Sepsis (Infections and infestations) | 7 | 6 | 7
Sepsis syndrome (Infections and infestations) | 1 | 0 | 0
Septic encephalopathy (Infections and infestations) | 0 | 1 | 0
Septic shock (Infections and infestations) | 0 | 3 | 3
Sinusitis (Infections and infestations) | 0 | 1 | 0
Staphylococcal bacteraemia (Infections and infestations) | 1 | 0 | 0
Staphylococcal infection (Infections and infestations) | 1 | 2 | 1
Streptococcal bacteraemia (Infections and infestations) | 1 | 0 | 0
Streptococcal sepsis (Infections and infestations) | 0 | 1 | 0
Subcutaneous abscess (Infections and infestations) | 1 | 0 | 0
Tonsillitis (Infections and infestations) | 1 | 0 | 1
Tooth infection (Infections and infestations) | 1 | 0 | 0
Tracheobronchitis (Infections and infestations) | 0 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 3 | 5 | 0
Urosepsis (Infections and infestations) | 2 | 3 | 2
Varicella (Infections and infestations) | 0 | 0 | 1
Vestibular neuronitis (Infections and infestations) | 1 | 0 | 0
Viral pericarditis (Infections and infestations) | 0 | 1 | 0
Vulval abscess (Infections and infestations) | 1 | 1 | 0
Wound infection (Infections and infestations) | 0 | 1 | 1
Accidental overdose (Injury, poisoning and procedural complications) | 1 | 1 | 0
Alcohol poisoning (Injury, poisoning and procedural complications) | 0 | 0 | 1
Anaesthetic complication pulmonary (Injury, poisoning and procedural complications) | 1 | 0 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 3 | 3
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Chest injury (Injury, poisoning and procedural complications) | 1 | 0 | 0
Concussion (Injury, poisoning and procedural complications) | 0 | 1 | 1
Craniocerebral injury (Injury, poisoning and procedural complications) | 1 | 0 | 1
Facial bones fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 3 | 3 | 0
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Femur fracture (Injury, poisoning and procedural complications) | 1 | 0 | 1
Fibula fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Foot fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Head injury (Injury, poisoning and procedural complications) | 0 | 1 | 0
Hip fracture (Injury, poisoning and procedural complications) | 2 | 1 | 1
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 2 | 4
Incarcerated incisional hernia (Injury, poisoning and procedural complications) | 1 | 0 | 0
Incisional hernia (Injury, poisoning and procedural complications) | 1 | 0 | 0
Intentional overdose (Injury, poisoning and procedural complications) | 1 | 0 | 0
Joint injury (Injury, poisoning and procedural complications) | 0 | 1 | 0
Laceration (Injury, poisoning and procedural complications) | 0 | 0 | 1
Lower limb fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1 | 0 | 1
Meniscus injury (Injury, poisoning and procedural complications) | 0 | 0 | 2
Near drowning (Injury, poisoning and procedural complications) | 1 | 0 | 0
Overdose (Injury, poisoning and procedural complications) | 2 | 0 | 0
Patella fracture (Injury, poisoning and procedural complications) | 2 | 0 | 0
Pelvic fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Pharyngeal injury (Injury, poisoning and procedural complications) | 0 | 1 | 0
Post procedural complication (Injury, poisoning and procedural complications) | 1 | 0 | 3
Post procedural discomfort (Injury, poisoning and procedural complications) | 0 | 0 | 1
Post procedural haematoma (Injury, poisoning and procedural complications) | 5 | 3 | 2
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 | 4 | 2
Post procedural inflammation (Injury, poisoning and procedural complications) | 1 | 0 | 0
Procedural intestinal perforation (Injury, poisoning and procedural complications) | 0 | 1 | 0
Procedural pain (Injury, poisoning and procedural complications) | 4 | 6 | 4
Rib fracture (Injury, poisoning and procedural complications) | 1 | 2 | 1
Road traffic accident (Injury, poisoning and procedural complications) | 1 | 1 | 1
Seroma (Injury, poisoning and procedural complications) | 1 | 0 | 0
Shunt malfunction (Injury, poisoning and procedural complications) | 1 | 0 | 0
Skin graft failure (Injury, poisoning and procedural complications) | 1 | 0 | 0
Spinal column injury (Injury, poisoning and procedural complications) | 0 | 1 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Spinal cord injury cervical (Injury, poisoning and procedural complications) | 1 | 0 | 0
Spinal fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Tendon rupture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Tibia fracture (Injury, poisoning and procedural complications) | 0 | 2 | 1
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 | 0 | 1
Traumatic haematoma (Injury, poisoning and procedural complications) | 1 | 0 | 0
Upper limb fracture (Injury, poisoning and procedural complications) | 1 | 0 | 1
Urinary retention postoperative (Injury, poisoning and procedural complications) | 0 | 0 | 1
Wound secretion (Injury, poisoning and procedural complications) | 1 | 0 | 0
Arthroscopy (Investigations) | 0 | 1 | 0
Blood bilirubin increased (Investigations) | 1 | 1 | 0
Blood creatine phosphokinase increased (Investigations) | 0 | 1 | 0
Blood creatinine increased (Investigations) | 0 | 1 | 0
Coronavirus test positive (Investigations) | 1 | 0 | 0
Fibrin D dimer increased (Investigations) | 1 | 0 | 0
Gamma-glutamyltransferase increased (Investigations) | 1 | 0 | 1
Haemoglobin decreased (Investigations) | 1 | 0 | 0
Human rhinovirus test positive (Investigations) | 0 | 1 | 0
Liver function test abnormal (Investigations) | 0 | 1 | 0
Red blood cell sedimentation rate increased (Investigations) | 0 | 1 | 0
Transaminases increased (Investigations) | 1 | 0 | 0
Troponin increased (Investigations) | 0 | 1 | 0
Weight increased (Investigations) | 0 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 1 | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 4 | 0
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 3 | 3 | 2
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 3 | 2 | 1
Electrolyte imbalance (Metabolism and nutrition disorders) | 1 | 0 | 0
Failure to thrive (Metabolism and nutrition disorders) | 0 | 1 | 0
Fluid overload (Metabolism and nutrition disorders) | 0 | 1 | 0
Gout (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypercreatininaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 2 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 1 | 2
Hypokalaemia (Metabolism and nutrition disorders) | 2 | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Lactic acidosis (Metabolism and nutrition disorders) | 0 | 0 | 1
Obesity (Metabolism and nutrition disorders) | 1 | 0 | 1
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 2
Arthritis (Musculoskeletal and connective tissue disorders) | 3 | 2 | 0
Bone disorder (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Costochondritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Fracture nonunion (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Gouty arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Inclusion body myositis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 2 | 0 | 2
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 3 | 3 | 6
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 | 1 | 2
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 3 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 2
Myopathy (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Myositis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 6 | 8 | 6
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Polymyalgia rheumatica (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Psoriatic arthropathy (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 3 | 0 | 1
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 | 0 | 1
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Tendon calcification (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Vertebral foraminal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2
Adenocarcinoma of salivary gland (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Anal squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 0
Benign hepatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Benign neoplasm of spinal cord (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Benign salivary gland neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Bladder transitional cell carcinoma recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Bone cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Brain neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 2 | 2
Breast cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Breast cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Cholangiocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Chronic lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Chronic myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Clear cell renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Colon adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Diffuse large B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 3
Endometrial adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1 | 0
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Endometrial cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Gastrointestinal stromal tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Glioblastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 1
Haemangiopericytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Hepatic cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Hepatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 8 | 6 | 3
Intraductal papillary mucinous neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Intraductal papilloma of breast (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Intraductal proliferative breast lesion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1 | 0
Invasive breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 | 0 | 2
Large intestine benign neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Lip and/or oral cavity cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 2 | 0
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 1
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Metastases to skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Neuroendocrine tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Oral papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2 | 1
Parathyroid tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Phaeochromocytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 0
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Pleomorphic adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 | 4 | 2
Prostate cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Prostate cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 2
Prostate cancer stage II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Renal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Squamous cell carcinoma of lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 0
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Tongue neoplasm malignant stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 2
Uterine leiomyosarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Ataxia (Nervous system disorders) | 1 | 0 | 0
Autonomic nervous system imbalance (Nervous system disorders) | 0 | 0 | 1
Brain mass (Nervous system disorders) | 0 | 1 | 0
Brain stem haemorrhage (Nervous system disorders) | 0 | 0 | 1
Carotid artery stenosis (Nervous system disorders) | 2 | 0 | 1
Cauda equina syndrome (Nervous system disorders) | 0 | 0 | 1
Cerebral haemorrhage (Nervous system disorders) | 0 | 0 | 1
Cerebral infarction (Nervous system disorders) | 0 | 0 | 1
Cerebral thrombosis (Nervous system disorders) | 0 | 0 | 1
Cerebrospinal fluid leakage (Nervous system disorders) | 1 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 1 | 3 | 1
Cervical radiculopathy (Nervous system disorders) | 0 | 0 | 2
Cognitive disorder (Nervous system disorders) | 1 | 0 | 1
Dementia (Nervous system disorders) | 1 | 0 | 0
Depressed level of consciousness (Nervous system disorders) | 0 | 1 | 0
Dizziness (Nervous system disorders) | 2 | 0 | 2
Dysarthria (Nervous system disorders) | 1 | 1 | 0
Encephalopathy (Nervous system disorders) | 1 | 0 | 1
Essential tremor (Nervous system disorders) | 0 | 1 | 0
Haemorrhage intracranial (Nervous system disorders) | 1 | 1 | 1
Headache (Nervous system disorders) | 1 | 1 | 0
Hemiparesis (Nervous system disorders) | 1 | 0 | 0
Hepatic encephalopathy (Nervous system disorders) | 1 | 2 | 0
Hypoaesthesia (Nervous system disorders) | 1 | 2 | 0
Intracranial aneurysm (Nervous system disorders) | 0 | 1 | 0
Intracranial pressure increased (Nervous system disorders) | 1 | 0 | 0
Ischaemic stroke (Nervous system disorders) | 1 | 3 | 1
Lacunar stroke (Nervous system disorders) | 1 | 0 | 0
Lumbosacral radiculopathy (Nervous system disorders) | 0 | 1 | 0
Metabolic encephalopathy (Nervous system disorders) | 0 | 1 | 0
Migraine (Nervous system disorders) | 1 | 4 | 1
Motor neurone disease (Nervous system disorders) | 1 | 0 | 0
Nerve compression (Nervous system disorders) | 1 | 0 | 0
Nervous system disorder (Nervous system disorders) | 0 | 0 | 1
Optic neuritis (Nervous system disorders) | 1 | 0 | 0
Parkinson's disease (Nervous system disorders) | 1 | 0 | 0
Parkinsonism (Nervous system disorders) | 1 | 0 | 0
Polyneuropathy (Nervous system disorders) | 1 | 0 | 0
Post herpetic neuralgia (Nervous system disorders) | 0 | 1 | 0
Presyncope (Nervous system disorders) | 0 | 3 | 0
Sciatica (Nervous system disorders) | 0 | 0 | 1
Seizure (Nervous system disorders) | 0 | 2 | 0
Sensory disturbance (Nervous system disorders) | 0 | 0 | 1
Spinal epidural haemorrhage (Nervous system disorders) | 1 | 0 | 0
Subarachnoid haemorrhage (Nervous system disorders) | 0 | 1 | 0
Syncope (Nervous system disorders) | 7 | 3 | 5
Thalamic infarction (Nervous system disorders) | 1 | 1 | 0
Transient global amnesia (Nervous system disorders) | 1 | 0 | 0
Transient ischaemic attack (Nervous system disorders) | 1 | 3 | 3
Trigeminal neuralgia (Nervous system disorders) | 1 | 0 | 0
VIIth nerve paralysis (Nervous system disorders) | 2 | 1 | 1
VIth nerve paralysis (Nervous system disorders) | 0 | 0 | 1
Vertebrobasilar insufficiency (Nervous system disorders) | 0 | 1 | 0
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 | 1 | 0
Adjustment disorder with depressed mood (Psychiatric disorders) | 1 | 0 | 0
Bipolar I disorder (Psychiatric disorders) | 0 | 1 | 2
Bipolar disorder (Psychiatric disorders) | 1 | 0 | 0
Completed suicide (Psychiatric disorders) | 1 | 0 | 2
Confusional state (Psychiatric disorders) | 0 | 2 | 1
Depression (Psychiatric disorders) | 3 | 0 | 1
Major depression (Psychiatric disorders) | 0 | 0 | 2
Mental disorder (Psychiatric disorders) | 0 | 1 | 1
Mental status changes (Psychiatric disorders) | 1 | 0 | 0
Panic disorder (Psychiatric disorders) | 0 | 1 | 0
Psychogenic seizure (Psychiatric disorders) | 1 | 1 | 1
Psychogenic tremor (Psychiatric disorders) | 0 | 0 | 1
Rapid eye movements sleep abnormal (Psychiatric disorders) | 1 | 0 | 0
Suicidal ideation (Psychiatric disorders) | 0 | 2 | 1
Suicide attempt (Psychiatric disorders) | 1 | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 6 | 13 | 4
Bladder prolapse (Renal and urinary disorders) | 0 | 0 | 1
Calculus ureteric (Renal and urinary disorders) | 2 | 1 | 1
Calculus urinary (Renal and urinary disorders) | 1 | 0 | 0
Cystitis haemorrhagic (Renal and urinary disorders) | 0 | 2 | 0
Diabetic nephropathy (Renal and urinary disorders) | 0 | 1 | 0
Hydronephrosis (Renal and urinary disorders) | 0 | 1 | 1
Lower urinary tract symptoms (Renal and urinary disorders) | 0 | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 5 | 5 | 5
Pelvi-ureteric obstruction (Renal and urinary disorders) | 0 | 0 | 1
Renal aneurysm (Renal and urinary disorders) | 1 | 0 | 0
Renal colic (Renal and urinary disorders) | 0 | 1 | 0
Renal failure (Renal and urinary disorders) | 1 | 0 | 0
Renal impairment (Renal and urinary disorders) | 0 | 1 | 0
Ureteric obstruction (Renal and urinary disorders) | 0 | 0 | 1
Urethral stenosis (Renal and urinary disorders) | 1 | 0 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 3 | 1 | 0
Breast haematoma (Reproductive system and breast disorders) | 1 | 0 | 0
Endometrial hyperplasia (Reproductive system and breast disorders) | 1 | 0 | 0
Endometrial thickening (Reproductive system and breast disorders) | 0 | 1 | 0
Menorrhagia (Reproductive system and breast disorders) | 1 | 1 | 0
Metrorrhagia (Reproductive system and breast disorders) | 0 | 0 | 1
Pelvic congestion (Reproductive system and breast disorders) | 1 | 0 | 0
Pelvic pain (Reproductive system and breast disorders) | 1 | 0 | 1
Pelvic prolapse (Reproductive system and breast disorders) | 0 | 1 | 0
Rectocele (Reproductive system and breast disorders) | 1 | 0 | 0
Uterine polyp (Reproductive system and breast disorders) | 0 | 1 | 0
Uterine prolapse (Reproductive system and breast disorders) | 0 | 1 | 0
Uterovaginal prolapse (Reproductive system and breast disorders) | 0 | 1 | 0
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 5 | 2
Asthma-chronic obstructive pulmonary disease overlap syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Bronchopneumopathy (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 5 | 3 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 5 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Idiopathic pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Nasopharyngeal polyp (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Organising pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pneumothorax spontaneous (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pulmonary alveolar haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 2
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pulmonary hilum mass (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 1
Angioedema (Skin and subcutaneous tissue disorders) | 0 | 2 | 0
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Dermatomyositis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Diabetic foot (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Hidradenitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Lichen sclerosus (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 5 | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Liver transplant (Surgical and medical procedures) | 2 | 1 | 1
Physiotherapy (Surgical and medical procedures) | 0 | 0 | 1
Rotator cuff repair (Surgical and medical procedures) | 0 | 0 | 1
ANXIETY-DEPRESSIVE DISORDER (Psychiatric disorders) | 1 | 0 | 0
INTRACRANIAL HEMORRHAGE (Injury, poisoning and procedural complications) | 1 | 0 | 0
PNEUMONIA METASTASIS OF OESOPHAGEAL CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Aortic dissection (Vascular disorders) | 0 | 1 | 0
Aortic stenosis (Vascular disorders) | 0 | 1 | 2
Arterial haemorrhage (Vascular disorders) | 0 | 1 | 0
Arterial occlusive disease (Vascular disorders) | 1 | 0 | 0
Arteriosclerosis (Vascular disorders) | 1 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 1 | 0
Hypertension (Vascular disorders) | 2 | 2 | 0
Hypertensive crisis (Vascular disorders) | 2 | 0 | 2
Hypertensive emergency (Vascular disorders) | 1 | 0 | 0
Hypotension (Vascular disorders) | 2 | 3 | 1
Orthostatic hypotension (Vascular disorders) | 1 | 1 | 0
Peripheral arterial occlusive disease (Vascular disorders) | 0 | 0 | 1
Shock (Vascular disorders) | 0 | 0 | 1
Shock haemorrhagic (Vascular disorders) | 0 | 2 | 0
Varicose vein (Vascular disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | OCA 10 Milligrams (mg) (N=825) | OCA 25 mg (N=827) | Placebo (N=825)
Pruritus (Skin and subcutaneous tissue disorders) | 294 | 470 | 210
Rash (Skin and subcutaneous tissue disorders) | 46 | 61 | 48
Pruritus generalised (Skin and subcutaneous tissue disorders) | 15 | 55 | 13
Urinary tract infection (Infections and infestations) | 147 | 151 | 133
Upper respiratory tract infection (Infections and infestations) | 88 | 103 | 84
Nasopharyngitis (Infections and infestations) | 82 | 80 | 70
Sinusitis (Infections and infestations) | 74 | 73 | 80
Bronchitis (Infections and infestations) | 81 | 66 | 66
Influenza (Infections and infestations) | 61 | 63 | 59
Nausea (Gastrointestinal disorders) | 148 | 165 | 150
Abdominal pain (Gastrointestinal disorders) | 139 | 135 | 132
Constipation (Gastrointestinal disorders) | 115 | 128 | 92
Abdominal pain upper (Gastrointestinal disorders) | 95 | 104 | 106
Diarrhoea (Gastrointestinal disorders) | 112 | 108 | 145
Vomiting (Gastrointestinal disorders) | 71 | 90 | 66
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 51 | 63 | 47
Abdominal distension (Gastrointestinal disorders) | 59 | 57 | 48
Dyspepsia (Gastrointestinal disorders) | 48 | 35 | 41
Low-density lipoprotein increased (Investigations) | 175 | 183 | 92
Blood cholesterol increased (Investigations) | 53 | 51 | 32
Blood creatinine increased (Investigations) | 53 | 43 | 43
Glycosylated haemoglobin increased (Investigations) | 47 | 40 | 37
Aspartate aminotransferase increased (Investigations) | 38 | 27 | 46
Alanine aminotransferase increased (Investigations) | 37 | 26 | 49
Gamma-glutamyltransferase increased (Investigations) | 28 | 14 | 43
Arthralgia (Musculoskeletal and connective tissue disorders) | 117 | 132 | 134
Back pain (Musculoskeletal and connective tissue disorders) | 136 | 105 | 120
Pain in extremity (Musculoskeletal and connective tissue disorders) | 67 | 67 | 66
Muscle spasms (Musculoskeletal and connective tissue disorders) | 47 | 49 | 60
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 65 | 53 | 61
Diabetes mellitus (Metabolism and nutrition disorders) | 112 | 99 | 94
Hyperlipidaemia (Metabolism and nutrition disorders) | 80 | 90 | 33
Hypercholesterolaemia (Metabolism and nutrition disorders) | 57 | 48 | 26
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 70 | 47 | 60
Fatigue (General disorders) | 148 | 135 | 138
Oedema peripheral (General disorders) | 47 | 39 | 42
Headache (Nervous system disorders) | 83 | 87 | 90
Dizziness (Nervous system disorders) | 62 | 53 | 55
Procedural pain (Injury, poisoning and procedural complications) | 58 | 50 | 44
Fall (Injury, poisoning and procedural complications) | 44 | 30 | 40
Cough (Respiratory, thoracic and mediastinal disorders) | 81 | 69 | 62
Insomnia (Psychiatric disorders) | 68 | 55 | 48
Depression (Psychiatric disorders) | 63 | 54 | 62
Anxiety (Psychiatric disorders) | 45 | 54 | 42
Cholelithiasis (Hepatobiliary disorders) | 50 | 66 | 30
Hypertension (Vascular disorders) | 106 | 97 | 88

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2021-05-04): https://cdn.clinicaltrials.gov/large-docs/51/NCT02548351/Prot_000.pdf
  • Statistical Analysis Plan (2023-01-31): https://cdn.clinicaltrials.gov/large-docs/51/NCT02548351/SAP_001.pdf